CLINICAL TRIAL: NCT02797717
Title: An International, Multicentre, Randomised Controlled Trial. Treatment for Classical Hodgkin Lymphoma in Children and Adolescents Standard Treatment (Chemotherapy and RT) Compared With Experimental Treatment (Chemotherapy Without RT or Restricted to RT)
Brief Title: Treatment for Classical Hodgkin Lymphoma in Children and Adolescents
Acronym: EuroNet-PHL-C2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GALIA AVRAHAMI (Other)
Collaborators: University of Giessen (Other)
Responsible Party: Sponsor-Investigator, GALIA AVRAHAMI, Senior pediatric oncologist physician, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: scmci160509ctil
Record Dates: First submitted 2016-04-12; First posted 2016-06-13 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Classical Hodgkins Lymphoma in Children and Adolescents.
MeSH Terms: interventions — Radiotherapy; Vincristine; Etoposide; Prednisone; Doxorubicin; Dacarbazine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A-"COPDAC-28" (Other): standard COPDAC-28 (chemotherapy cycle:Cyclophosphamide,Doxorubicin,Prednisone,Dacarbazine), chemotherapy and standard involved node radiotherapy.
  drugs: Prednisone 40mg/m2/day,P.O,day 1-day 15. Dacarbazine 250mg/m2, I.V. , infusion,day 1- day 3. Vincristine 15mg/m2 , I.V. , day1+day 8. Cyclophosphamide 500mg/m2,infusion,day 1+day 8.
  Interventions: Radiation: Radiotherapy:; Drug: Vincristine; Drug: Prednisone; Drug: Dacarbazine; Drug: Cyclophosphamide
- B- "DECOPDAC-21" (Experimental): DECOPDAC-21(chemotherapy cycle:Dacarbazine,Etoposide,Doxorubicin,Cyclophosphamide,Prednisone,Vincristine) intensified chemotherapy and no RT or restricted fields of radiotherapy.
  Drugs: Prednisone 40mg/m2/day,P.O,day 1-day 15:
  Dacarbazine 250mg/m2, I.V. , infusion,day 1- day 3 Vincristine 15mg/m2 , I.V. , day1+day 8 Cyclophosphamide 625mg/m2,infusion,day1+day2 Etoposide 100mg/m2/day,infusion,day 1- day 3 Doxorubicin 25mg/m2, infusion, day 1
  Interventions: Radiation: Radiotherapy:; Drug: Vincristine; Drug: Etoposide; Drug: Prednisone; Drug: Doxorubicin; Drug: Dacarbazine; Drug: Cyclophosphamide

INTERVENTIONS:
Radiation: Radiotherapy: — All patients will have 2 "OPEA"cycles(chemotherapy cycle:Vincristine,Etoposide,Prednisone,doxorubicin) ,After assignment ( by randomization) to one of the arms the patient will be treated accordingly . response assessment will be done after "OPEA" cycles (ERA) and after cycles of "copdac 28" or DECOPDAC 21(LRA).according to the assessments results patients will have radiotherapy or not.
Drug: Vincristine — ARM A and ARM B
Drug: Etoposide — ARM B , 100mg/m2/day
  Arms: B- "DECOPDAC-21"
Drug: Prednisone — ARM A and ARM B , 40mg/m2/day p.o
Drug: Doxorubicin — ARM B , 25mg/m2
  Arms: B- "DECOPDAC-21"
Drug: Dacarbazine — ARM A and ARM B , 250mg/m2 i.v
Drug: Cyclophosphamide — ARM A and ARM B , 625mg/m2 i.v

SUMMARY:
Reduction of the indication for radiotherapy (RT) in newly diagnosed patients with classical Hodgkins lymphoma without compromising cure rates. Investigation of a chemotherapy intensification randomisation in intermediate and advanced classical Hodgkins lymphoma patients to compensate for reduction in RT.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed primary diagnosis of classical Hodgkin's lymphoma.
2. patients under 18 years of age on the date of written informed consent. In specialized Teenage and Young Adult (TYA) units in Australia, France, Italy, New Zealand and United Kingdom patients up to under 25 years of age can also be enrolled. Lower age limits will be country specific according to national laws or formal insurance requirements that may preclude very young patients.
3. written informed consent of the patient and/or the patient's parents or guardian according to national laws.
4. negative pregnancy test within 2 weeks prior to starting treatment for female patients with childbearing potential

Exclusion Criteria: (Patients with one or more of the following criterion are excluded)

1. prior chemotherapy or radiotherapy for other malignancies
2. pre-treatment of Hodgkin's lymphoma (except for steroid pre-phase to a maximum of 7-10 days for emergency treatment of a large mediastinal tumour).
3. diagnosis of lymphocyte-predominant Hodgkin's lymphoma
4. other (simultaneous) malignancies
5. contraindication or known hypersensitivity to study drugs
6. severe concomitant diseases (e.g. immune deficiency syndrome)
7. known HIV-positivity
8. residence outside the participating countries where long term follow-up cannot be guaranteed
9. pregnancy and / or lactation
10. patients who are sexually active and are unwilling to use adequate contraception during therapy and for one month after last trial treatment
11. current or recent (within 30 days prior to date of written informed consent) treatment with another investigational drug or participation in another interventional clinical trial

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2200 (Estimated)
Dates: Start 2015-11; Primary Completion 2022-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Increase event free survival rate from 88% to 93% | Will be assessed once a year up to 5 years after end of treatment.
  Methods of measurement: chest X-ray; US neck, abdomen and pelvis; lung function; T4,Throid Stimulating Hormone ,US of thyroid; MRI of initially involved region; chest CT in patients with initial lung involvement.

SECONDARY OUTCOMES:
comparison of haematotoxicity between arm A and arm B | Will be assessed in day 0,day 8,day 11,day 17 and day 21 of each cycle
  Evaluation of haematotoxicity by documentation of blood count courses during "OEPA", COPDAC-28 and DECOPDAC-21 cycles. Comparison between COPDAC-28 versus DECOPDAC-21.
  For ERA(early response assessment) PET(Positron Emission Tomography)-positive patients to compare to the LRA (late response assessment)PET-positivity rates after consolidation chemotherapy with COPDAC-28 or DECOPDAC-21.

CONTACTS AND LOCATIONS:
Overall Officials: Dieter K.rholz, Prof. Dr., Study Chair — Universit.tsklinikum Giessen; Galia Avrahami, MD, Principal Investigator — Schneider children medical center,Kaplan 14 Petach-Tikva,Israel
Locations (1):
- Schneider children's medical center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No